CLINICAL TRIAL: NCT02561273
Title: A Phase I/II Trial of CHOEP Chemotherapy Plus Lenalidomide as Front Line Therapy for Patients With Stage II, III and IV Peripheral T-Cell Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy & Lenalidomide in Newly Diagnosed Stage II-IV Peripheral T-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0511-14-FB; NCI-2015-00088 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RV-CL-PTCL-PI-003858 (Other Grant/Funding Number: Celgene Corporation); P30CA036727 (NIH)
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Negative; Anaplastic Large Cell Lymphoma, ALK-Positive; Hepatosplenic T-Cell Lymphoma; Peripheral T-Cell Lymphoma, Not Otherwise Specified; Stage II Angioimmunoblastic T-cell Lymphoma; Stage II Enteropathy-Associated T-Cell Lymphoma; Stage III Angioimmunoblastic T-cell Lymphoma; Stage III Enteropathy-Associated T-Cell Lymphoma; Stage IV Angioimmunoblastic T-cell Lymphoma; Stage IV Enteropathy-Associated T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Enteropathy-Associated T-Cell Lymphoma | interventions — Cyclophosphamide; Doxorubicin; Etoposide; Lenalidomide; Peripheral Blood Stem Cell Transplantation; Prednisone; deltacortene; prednylidene; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (combination chemotherapy, lenalidomide) (Experimental): Patients receive cyclophosphamide IV, doxorubicin hydrochloride IV and vincristine sulfate IV on day 1, etoposide IV over 30-60 minutes on days 1-3, prednisone PO on days 1-5, and lenalidomide PO on days 1-10. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients responding after 6 courses of treatment may then undergo an autologous stem cell transplant or receive maintenance lenalidomide at the discretion of the physician or patient choice as follows:
  TRANSPLANT: Patients undergo autologous stem cell transplant per standard of care.
  MAINTENANCE LENALIDOMIDE: Patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Prednisone; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous stem cell transplant
  Other Names: Autologous Stem Cell Transplantation
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo peripheral blood stem cell transplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide when given together with combination chemotherapy and to see how well they work in treating patients with newly diagnosed stage II-IV peripheral T-cell non-Hodgkin's lymphoma. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Lenalidomide may stop the growth of peripheral T-cell non-Hodgkin's lymphoma by blocking the growth of new blood vessels necessary for cancer growth. Giving combination chemotherapy with lenalidomide may be a better treatment for peripheral T-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and efficacy of lenalidomide in combination with standard induction therapy (CHOEP- cyclophosphamide, doxorubicin [doxorubicin hydrochloride], etoposide, vincristine [vincristine sulfate] and prednisone) in patients with newly diagnosed stage II, III and IV peripheral T-cell lymphoma not otherwise specified (NOS), anaplastic large cell lymphoma (anaplastic lymphoma receptor tyrosine kinase [ALK] negative) (ALK positive if International Prognostic Index [IPI] 3, 4, or 5), angioimmunoblastic T-cell lymphoma, enteropathy associated T-cell lymphoma or hepatosplenic gamma delta T-cell lymphoma.

II. To establish the maximum tolerated dose of lenalidomide in combination with CHOEP chemotherapy. (Phase I) III. To assess the efficacy (complete response rate) of this combination. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate overall response rate (complete response [CR] + partial response [PR]) of the combination of lenalidomide and CHOEP chemotherapy.

II. To evaluate the safety and tolerability of the regimen. III. To assess the 2 year progression free survival (PFS) and overall survival (OS) using this regimen.

OUTLINE: This is a phase I, dose-escalation study of lenalidomide, followed by a phase II study.

Patients receive cyclophosphamide intravenously (IV), doxorubicin hydrochloride IV and vincristine sulfate IV on day 1, etoposide IV over 30-60 minutes on days 1-3, prednisone orally (PO) on days 1-5, and lenalidomide PO on days 1-10. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients responding after 6 courses of treatment may then undergo an autologous stem cell transplant or receive maintenance lenalidomide at the discretion of the physician or patient choice as follows:

TRANSPLANT: Patients undergo autologous stem cell transplant per standard of care.

MAINTENANCE LENALIDOMIDE: Patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed new diagnosis of stage II, III and IV peripheral T-cell non-Hodgkin's lymphoma not otherwise specified (NOS), anaplastic large cell lymphoma (ALK negative) (ALK positive if IPI 3, 4, or 5), angioimmunoblastic T-cell lymphoma, enteropathy associated T-cell lymphoma, hepatosplenic gamma delta T-cell lymphoma
* Pathology material: hematoxylin and eosin (H&E) stain and immunohistochemistry (IHC) slides or a representative formalin-fixed paraffin-embedded (FFPE) tissue block along with the pathology report from initial diagnosis, should be sent to be reviewed, and the diagnosis confirmed by Mayo Clinic department (retrospective diagnostic review: treatment may commence prior to the Mayo Clinic review)
* No prior therapy with the exception of prior radiation therapy and/or prednisone alone, at the discretion of the investigator based on current diagnosis and clinical condition; this prednisone treatment will not count toward the 6 cycles of treatment given in the study
* Expected survival duration of > 3 months
* Karnofsky performance status > 70
* Absolute neutrophil count (ANC) > 1000 cells/mm^3, unless cytopenias due to non-Hodgkin lymphoma (NHL) (i.e., bone marrow involvement or splenomegaly)
* Platelet count > 100,000/uL or > 75,000/uL if bone marrow (BM) involvement or splenomegaly
* Total bilirubin =< 1.5 x upper normal limit, or =< 3 x upper normal limit if documented hepatic involvement with lymphoma, or =< 5 x upper normal limit if history of Gilbert's disease
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper normal limit (=< 5 x upper normal limit if documented hepatic involvement with lymphoma)
* Serum creatinine < 2.0 mg/dL or calculated creatinine clearance (CrCl) > 45 mL/min (Cockcroft-Gault)
* Prothrombin time (PT) or international normalized ratio (INR), and partial thromboplastin time (PTT) =< 1.5 x upper limit of normal unless patient is receiving anticoagulants; if patient is on warfarin therapy, levels should be within therapeutic range
* If currently not on anticoagulation medication, willing and able to take aspirin (81 or 325 mg) daily; if aspirin is contraindicated, the patient may be considered for the study if on therapeutic dose warfarin or low molecular weight heparin; patients unable to take any prophylaxis are not eligible
* Patients with measurable disease; patients with non-measurable but evaluable disease may be eligible after discussion with the principal investigator (PI); baseline measurements and evaluations must be obtained within 6 weeks of registration to the study; abnormal positron emission tomography (PET)/computed tomography (CT) scans will not constitute evaluable disease, unless verified by CT scan or other appropriate imaging
* Patients with measurable disease must have at least one objective measurable disease parameter; a clearly defined, bi-dimensionally measurable defect or mass measuring at least 1.5 cm in diameter on the CT portion of a PET/CT or CT scan or magnetic resonance imaging (MRI) (if appropriate) will constitute measurable disease; proof of lymphoma in the liver is required by a confirmation biopsy; skin lesions can be used as measurable disease provided bi-dimensional measurements are possible
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of the REMS program
* Women must not be pregnant or breast-feeding

  * Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program
  * All females of childbearing potential must have a blood test within 2 weeks prior to registration to rule out pregnancy
  * Pregnancy testing is not required for post-menopausal or surgically sterilized women
* Male and female patients of reproductive potential must agree follow accepted birth control measures
* Patient must be able to adhere to the study visit schedule and other protocol requirements
* Patients must be willing to give written informed consent, and sign an institutionally approved consent form before performance of any study-related procedure not part of normal medical care as noted above; with the exception of 1 cycle of chemotherapy based on current diagnosis and clinical condition, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* No serious disease or condition that, in the opinion of the investigator, would compromise the patient's ability to participate in the study

Exclusion Criteria:

* Pregnant or breast feeding females
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); patients who are seropositive ( i.e. hepatitis B core antibody positive; quantitative deoxyribonucleic acid [DNA] negative) are eligible with appropriate prophylaxis
* Major surgery within 2 weeks of study drug administration
* Prior malignancies within the past 3 years with exception of adequately treated basal cell, squamous cell skin cancer, or thyroid cancer; carcinoma in situ of the cervix or breast; prostate cancer of Gleason grade 6 or less with stable prostate-specific antigen (PSA) levels
* Patients with a diagnosis of other peripheral T-cell lymphoma (PTCL) histologies other than those specified in the inclusion criteria
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, or antiviral drugs
* Any other clinically significant medical disease or condition laboratory abnormality or psychiatric illness that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
* Known hypersensitivity to thalidomide or lenalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, lenalidomide or similar drugs
* Ejection fraction of < 45% by either multi gated acquisition scan (MUGA) or echocardiogram (ECHO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Lunning, Principal Investigator — University of Nebraska
Locations (8):
- United States (8):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of Colorado Cancer Center, Anschutz Cancer Pavilion, Aurora, Colorado
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per the protocol, date of enrollment is defined as the date of consent. For this study 54 participants were consented. 10 were determined to be ineligible and not assigned to a study group.
Groups:
- 10 mg Lenalidomide Participants; 15 mg Lenalidomide Participants: Patients receive cyclophosphamide IV, doxorubicin hydrochloride IV and vincristine sulfate IV on day 1, etoposide IV over 30-60 minutes on days 1-3, prednisone PO on days 1-5, and lenalidomide PO on days 1-10. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients responding after 6 courses of treatment may then undergo an autologous stem cell transplant or receive maintenance lenalidomide at the discretion of the physician or patient choice as follows:
  TRANSPLANT: Patients undergo autologous stem cell transplant per standard of care.
  MAINTENANCE LENALIDOMIDE: Patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous stem cell transplant
Period: Overall Study
Arm/Group | 10 mg Lenalidomide Participants | 15 mg Lenalidomide Participants
Started | 40 | 4
Completed | 39 | 4
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg Lenalidomide Participants | 15 mg Lenalidomide Participants | Total
Number analyzed (Participants) | 39 | 4 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13) | 62 (4) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 2 | 21
  Male | 20 | 2 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 30 | 2 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 39 | 4 | 43

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Lenalidomide and CHOEP
Description: MTD is defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients) (Phase I) within the first cycle of study treatment.
Time Frame: 21 days
Population: Eight subjects were dosed at 10 mg dose and 4 subjects were dosed at 15 mg dose.
Measure: Number; unit: milligrams
Groups:
- Treatment (Combination Chemotherapy, Lenalidomide): Patients receive cyclophosphamide IV, doxorubicin hydrochloride IV and vincristine sulfate IV on day 1, etoposide IV over 30-60 minutes on days 1-3, prednisone PO on days 1-5, and lenalidomide PO on days 1-10. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients responding after 6 courses of treatment may then undergo an autologous stem cell transplant or receive maintenance lenalidomide at the discretion of the physician or patient choice as follows:
  TRANSPLANT: Patients undergo autologous stem cell transplant per standard of care.
  MAINTENANCE LENALIDOMIDE: Patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous stem cell transplant
Arm/Group | Treatment (Combination Chemotherapy, Lenalidomide)
Number analyzed (Participants) | 12
milligrams | 10

2. Primary Outcome: Number of Participants With Adverse Events Graded According to Common Toxicity Criteria (CTC) (Phase I)
Description: Non-hematologic toxicities will be evaluated via the ordinal CTC standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by dose level and patient will be explored and summarized.
Time Frame: Up to 6 cycles of treatment (approximately 5 months)
Population: Toxicity was measured for all subjects dosed during Phase 1 of the study. 10 mg and 15 mg dose levels.
Measure: Count of Participants; unit: Participants
Groups:
- 10 mg Lenalidomide Participants; 15 mg Lenalidomide Participants: Patients receive cyclophosphamide IV, doxorubicin hydrochloride IV and vincristine sulfate IV on day 1, etoposide IV over 30-60 minutes on days 1-3, prednisone PO on days 1-5, and lenalidomide PO on days 1-10. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients responding after 6 courses of treatment may then undergo an autologous stem cell transplant or receive maintenance lenalidomide at the discretion of the physician or patient choice as follows:
  TRANSPLANT: Patients undergo autologous stem cell transplant per standard of care.
  MAINTENANCE LENALIDOMIDE: Patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | 10 mg Lenalidomide Participants | 15 mg Lenalidomide Participants
Number analyzed (Participants) | 8 | 4
Participants
  grade 3,4 neutropenia | 5 | 4
  grade 3, 4 anemia | 3 | 3
  grade 3, 4 thrombocytopenia | 2 | 3
  grade 3,4 neutropenia fever | 4 | 0
  grade 3, 4 diarrhea | 0 | 2
  grade 3, 4 hyperglycemia | 0 | 2
  grade 3, 4 hypokalemia | 0 | 1
  grade 3, 4 hypotension | 0 | 1
  grade 3, 4 hyperbilirubinemia | 0 | 1
  grade 3, 4 mucositis | 0 | 2
  grade 3,4 nausea | 0 | 2
  grade 3,4 vomiting | 0 | 1

3. Primary Outcome: Complete Response Rate (Phase II)
Description: A success is defined to be an objective status of CR after completion of 6 cycles of treatment. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. A 95% confidence interval for the true overall CR rate will be calculated according to the method of Duffy and Santner.
Time Frame: Up to the completion of course 6 (18 weeks)
Population: Assessment based on phase II patients given the maximum tolerated dose level (10 mg) as the Intent to treat (ITT) group of subjects. 39 subjects were dosed with 10 mg dose of Lenalidamide as the ITT group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (Combination Chemotherapy, Lenalidomide): Patients receive cyclophosphamide IV, doxorubicin hydrochloride IV and vincristine sulfate IV on day 1, etoposide IV over 30-60 minutes on days 1-3, prednisone PO on days 1-5, and lenalidomide PO on days 1-10. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients responding after 6 courses of treatment may then undergo an autologous stem cell transplant or receive maintenance lenalidomide at the discretion of the physician or patient choice as follows:
  TRANSPLANT: Patients undergo autologous stem cell transplant per standard of care.
  MAINTENANCE LENALIDOMIDE: Patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous stem cell transplant
  Cyclophosphamide: Given IV
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo peripheral blood stem cell transplant
  Prednisone: Given PO
  Vincristine Sulfate: Given IV
Arm/Group | Treatment (Combination Chemotherapy, Lenalidomide)
Number analyzed (Participants) | 39
percentage of participants | 49 [33 to 64]

4. Primary Outcome: Overall Response Rate
Description: The ORR will be estimated by the total number of patients who achieve a PR or CR at the end of six cycles of treatment divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true ORR will be calculated.
Time Frame: Up to the completion of course 6 (18 weeks)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Combination Chemotherapy, Lenalidomide)
Number analyzed (Participants) | 39
percentage of participants | 69 [54 to 81]

5. Secondary Outcome: Number of Participants With Adverse Events Graded According to CTC (Phase II)
Description: The toxicity profile will be further assessed based on phase II patients. Overall toxicity incidence of maximum tolerated dose level of the Intent to treat (ITT) group of subjects is summarized.
  39 subjects were dosed with 10 mg dose of Lenalidamide as the ITT group.
Time Frame: Up to 1 year
Population: Safety data for the Intent to treat (ITT) group of subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Combination Chemotherapy, Lenalidomide)
Number analyzed (Participants) | 39
Participants
  grade 3,4 neutropenia | 27
  grade 3, 4 leukopenia | 25
  grade 3, 4 anemia | 17
  grade 3, 4 thrombocytopenia | 17
  grade 3, 4 lymphopenia | 18
  grade 3, 4 febrile neutropenia | 15
  grade 3, 4 diarrhea | 3
  grade 3, 4 Peripheral sensory neuropathy | 2
  grade 3, 4 fatigue | 1
  grade 3, 4 nausea | 1
  grade 3, 4 anorexia | 1
  grade 3, 4 vomiting | 1
  grade 3, 4 mucositis oral | 1
  grade 3, 4 Rash maculo-papular | 1
  grade 3, 4 hypotension | 1
  grade 3, 4 back pain | 1

6. Secondary Outcome: Overall Survival
Description: The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause, assessed up to 1 year
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Combination Chemotherapy, Lenalidomide)
Number analyzed (Participants) | 39
percentage of participants | 89 [74 to 96]

7. Secondary Outcome: Progression-free Survival
Description: The distribution of PFS will be estimated using the method of Kaplan-Meier. The PFS rate at 2 years will be estimated. A 2-year PFS rate of 60% will be considered of interest.
Time Frame: Time from registration to progression or death due to any cause, assessed up to 2 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Combination Chemotherapy, Lenalidomide)
Number analyzed (Participants) | 39
percentage of participants | 55 [37 to 70]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent until 30 days post after the last administration of study drug (lenalidomide). For subjects going on to transplant after Len-CHOEP treatment this was approximately 5 months. For subjects going on the the maintenance len treatment instead of transplant upto an additional 1 year of maintenance lenalidomide treatment was allowed. (17 months total)
Groups:
- Treatment (10 mg Lenalidomide); Treatment (15 mg Lenalidomide): Patients receive cyclophosphamide IV, doxorubicin hydrochloride IV and vincristine sulfate IV on day 1, etoposide IV over 30-60 minutes on days 1-3, prednisone PO on days 1-5, and lenalidomide PO on days 1-10. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients responding after 6 courses of treatment may then undergo an autologous stem cell transplant or receive maintenance lenalidomide at the discretion of the physician or patient choice as follows:
  TRANSPLANT: Patients undergo autologous stem cell transplant per standard of care.
  MAINTENANCE LENALIDOMIDE: Patients receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous stem cell transplant
Arm/Group | Treatment (10 mg Lenalidomide) | Treatment (15 mg Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 9/39 | 1/4
Serious Adverse Events (participants affected / at risk) | 14/39 | 2/4
Other Adverse Events (participants affected / at risk) | 32/39 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (10 mg Lenalidomide) (N=39) | Treatment (15 mg Lenalidomide) (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 1
platelet count decreased (Blood and lymphatic system disorders) | 7 | 0
Neutrophil count decreased (Blood and lymphatic system disorders) | 5 | 1
fever (General disorders) | 5 | 0
anemia (Blood and lymphatic system disorders) | 5 | 0
sepsis (Infections and infestations) | 5 | 0
diarrhea (Gastrointestinal disorders) | 2 | 1
hypotension (Vascular disorders) | 2 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
White blood cells decreased (Blood and lymphatic system disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
cardiac arrest (Cardiac disorders) | 1 | 0
colitis (Gastrointestinal disorders) | 1 | 0
creatinine increased (Investigations) | 1 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
fatigue (General disorders) | 1 | 0
gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
T3 ADRENAL CORTICAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
dizziness (Nervous system disorders) | 0 | 1
gait disturbance (General disorders) | 0 | 1
hearing impaired (Ear and labyrinth disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 0 | 1
ACUTE ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (10 mg Lenalidomide) (N=39) | Treatment (15 mg Lenalidomide) (N=4)
Fatigue (General disorders) | 32 | 4
White blood cell decreased (Investigations) | 26 | 3
Neutrophil count decreased (Investigations) | 25 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 2
Anemia (Blood and lymphatic system disorders) | 23 | 3
Lymphocyte count decreased (Investigations) | 20 | 4
Platelet count decreased (Investigations) | 18 | 3
Nausea (Gastrointestinal disorders) | 17 | 2
diarrhea (Gastrointestinal disorders) | 16 | 2
peripheral sensory neuropathy (Nervous system disorders) | 16 | 1
constipation (Gastrointestinal disorders) | 13 | 1
dizziness (Nervous system disorders) | 11 | 0
Anorexia (Gastrointestinal disorders) | 10 | 0
mucositis, oral (Gastrointestinal disorders) | 10 | 2
Vomiting (Gastrointestinal disorders) | 10 | 1
rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3
hypotension (Vascular disorders) | 8 | 1
infections and infestation, Other (Infections and infestations) | 8 | 1
general disorders -Other (General disorders) | 7 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0
back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Anxiety (Psychiatric disorders) | 5 | 0
dysgeusia (Nervous system disorders) | 5 | 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
headache (Nervous system disorders) | 5 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 | 0
weight loss (Investigations) | 5 | 0
chills (General disorders) | 4 | 1
fever (General disorders) | 4 | 1
other gastrointestinal disorders (Gastrointestinal disorders) | 4 | 0
malaise (General disorders) | 4 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 4 | 0
pain (General disorders) | 4 | 2
syncope (Nervous system disorders) | 4 | 0
Other blood and lymphatic disorders (Blood and lymphatic system disorders) | 3 | 0
dry eye (Eye disorders) | 3 | 0
dysphagia (Gastrointestinal disorders) | 3 | 0
edema limbs (General disorders) | 3 | 1
hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1
hypokalemia (Metabolism and nutrition disorders) | 3 | 1
hyponatremia (Metabolism and nutrition disorders) | 3 | 1
Infusion related reaction (General disorders) | 3 | 0
other nervous system disorders (Nervous system disorders) | 3 | 0
other respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 | 1
sinus tachycardia (Cardiac disorders) | 3 | 0
sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0
blood bilirubin increased (Investigations) | 2 | 1
dehydration (Metabolism and nutrition disorders) | 2 | 0
external ear inflammation (Ear and labyrinth disorders) | 2 | 0
fall (Injury, poisoning and procedural complications) | 2 | 0
gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
hypertension (Vascular disorders) | 2 | 0
hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
insomnia (Psychiatric disorders) | 2 | 0
lymphedema (Vascular disorders) | 2 | 0
other musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 | 0
pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0
peripheral motor neuropathy (Nervous system disorders) | 2 | 0
rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
urinary frequency (Renal and urinary disorders) | 2 | 0
urinary tract infection (Infections and infestations) | 2 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
blurred vision (Eye disorders) | 0 | 1
creatinine increased (Investigations) | 0 | 1
dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
non-cardiac chest pain (General disorders) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
DRAINAGE FROM BIOPSY SITE (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT02561273/Prot_SAP_000.pdf